CLINICAL TRIAL: NCT05006066
Title: The Effect of the Nature And Frequency of a Stimulation on the Amplitude of the Temporal Summation of Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022-4323
Record Dates: First submitted 2021-07-21; First posted 2021-08-16 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Healthy
Keywords: Temporal Summation; Mechanical Stimulation; Heat Pain Stimulation; Thermode
MeSH Terms: interventions — Postsynaptic Potential Summation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy volunteers - Pain-Free: Each participant will be stimulated with 4 temporal summation stimulation conditions:
  * continuous thermal (1 stimulation of two minutes)
  * repetitive thermal (30 stimulations of 1 second)
  * continuous mechanical (1 stimulation of two minutes)
  * repetitive mechanical (30 stimulation of 1 second)
  Interventions: Other: Temporal Summation

INTERVENTIONS:
Other: Temporal Summation — 4 type of stimulations applied on the right arm

SUMMARY:
Temporal summation is a mechanism that enhances pain perception. It is a natural mechanism present in most individuals. Generally, temporal summation is measured by the application of a moderately painful stimulation for several seconds.However, there is still no official recommendation in the literature. There is therefore a great disparity in the protocols. Some studies apply thermal stimulation (heating the skin) while others apply mechanical stimulation (applying pressure). Another point of contention is that some studies apply continuous stimulation for 2 minutes while others apply a series of several small stimulation of 1 second). Between these studies, the amplitude of temporal summation varies according to the stimulation performed. Note also that the study population is also very different between studies. In these conditions, it remains difficult to know the impact of the nature of the stimulation on the measured amplitude of the temporal summation.

DETAILED DESCRIPTION:
Objective: To determine the effect of the nature and frequency of the stimulation used to measure one of the physiological mechanisms of pain

Methods: In order to meet the objective, 34 pain-free participants will be recruited (17 females and 17 males) between the ages of 18 and 30 years. A single visit will be proposed (approximately 1 h). Each participant will be stimulated with 4 stimulation conditions:

* continuous thermal (1 stimulation of two minutes)
* repetitive thermal (30 stimulations of 1 second)
* continuous mechanical (1 stimulation of two minutes)
* repetitive mechanical (30 stimulation of 1 second) In order to control certain psychological parameters, questionnaires measuring anxiety, depression and fear of pain will be administered. This will allow the investigation team to perform subgroup analyses if necessary. A repeated measures analysis of variance will be performed to meet the objective.

Anticipated Results: The objective of this project is to determine the impact of different stimuli on the measurement of a pain mechanism. In this sense, the results will be important since they will allow to develop recommendations to optimize the measurement of this mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 to 30 years, able to consent (understand English or French)
* No chronic pain
* No primary sensory disorders

Exclusion Criteria:

* Presence of upper extremity injuries
* Absence of anxiety symptoms (HADs Score < 6) (Appendix 1)
* Presence of cardiovascular disease / neurocognitive disorders / mental illness
* Pregnant or postpartum women less than one year old

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: For this project, healthy males and females (1:1 ratio) between the ages of 18 and 30 will represent our target population
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Temporal Summation of Pain - repetitive thermal stimulation | During stimulation
  Temporal Summation of pain referred to the change of pain perception during a painful stimulation. Temporal summation will be calculated by the difference in pain perception (on a 0-100 scale) and the beginning and at the end of each stimulation sequence. Temporal summation will be express as a percentage of increased.
Temporal Summation of Pain - continuous thermal stimulation | During stimulation
  Temporal Summation of pain referred to the change of pain perception during a painful stimulation. Temporal summation will be calculated by the difference in pain perception (on a 0-100 scale) and the beginning and at the end of each stimulation sequence. Temporal summation will be express as a percentage of increased.
Temporal Summation of Pain - continuous mechanical stimulation | During stimulation
  Temporal Summation of pain referred to the change of pain perception during a painful stimulation. Temporal summation will be calculated by the difference in pain perception (on a 0-100 scale) and the beginning and at the end of each stimulation sequence. Temporal summation will be express as a percentage of increased.
Temporal Summation of Pain - repetitive mechanical stimulation | During stimulation
  Temporal Summation of pain referred to the change of pain perception during a painful stimulation. Temporal summation will be calculated by the difference in pain perception (on a 0-100 scale) and the beginning and at the end of each stimulation sequence. Temporal summation will be express as a percentage of increased.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Léonard, Ph.D, Principal Investigator — Université de Sherbrooke
Locations (1):
- Université de Sherbrooke, Sherbrooke, Quebec, Canada